CLINICAL TRIAL: NCT06808321
Title: Evaluation of Clinical Outcomes of Benidipine in Hypertensive and/or Chronic Coronary Syndrome Patients in the Turkish Population
Brief Title: Benidipine in Hypertensive and/or Chronic Coronary Syndrome Patients
Acronym: Benidipine-TR
Status: Enrolling by invitation | Type: Observational
Sponsor: The Society of Prevention and Awareness of Cardiovascular Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-01
Record Dates: First submitted 2025-01-26; First posted 2025-02-05 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Chronic Coronary Syndrome; Hypertension; Angina Pectoris
Keywords: Coronary artery disease; Hypertension; Angina pectoris
MeSH Terms: conditions — Hypertension; Angina Pectoris; Coronary Artery Disease | interventions — benidipine hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Benidipine Hydrochloride — The safety and efficacy of a dihydropyridine calcium channel blocker for the treatment of high blood pressure and/or angina pectoris

SUMMARY:
Evaluation of the clinical outcomes of Benidipine initiated by physician's preference in patients with hypertension and/or angina pectoris (chronic coronary syndrome) presenting to cardiology outpatient clinics in Turkey.

DETAILED DESCRIPTION:
* Benidipine is a dihydropyridine calcium channel blocker used in the treatment of hypertension and angina pectoris. There are currently no large-scale observational studies in these patient groups in Turkey.
* There is no record of benidipine in clinicaltrials.gov, which is an important database especially for the registration of drug and interventional studies.
* Therefore, it will be extremely important to include this study in clinicaltrials.gov and to evaluate the clinical efficacy of Bendipine in patients with hypertensive and/or angina pectoris in 7 geographical regions of Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertension and/or angina pectoris on the background of chronic coronary syndrome who have been receiving Benidipine treatment for at least 1 month and will continue to receive Benidipine treatment
* Male or female outpatients, 18-80 years of age
* Patients with mild to moderate essential hypertension who have been receiving or will continue Benidipine treatment for at least 1 month
* Outpatients with clinically stable angina pectoris and patients who have been receiving or will continue Benidipine treatment for at least 1 month
* Those who signed the written informed consent form

Exclusion Criteria:

* Patients with secondary hypertension
* Emergency hypertensive patients
* Having to take other medications during the study that may affect blood pressure
* Allergic to DHP calcium antagonists
* Evidence of decompensated congestive heart failure, unstable angina or severe arrhythmia
* Severe renal or hepatic dysfunction
* Pregnant or lactating women
* Participation in other clinical trials within 3 months prior to this study
* Patients who did not sign the consent form of the study

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting to cardiology outpatient clinics in Turkey with hypertension and/or angina pectoris (chronic coronary syndrome)
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The Percentage of Patients Achieving Target Sitting Blood Pressure of Less Than 130/85 | 3 months
Change in angina symptom severity as measured by the Seattle Angina Questionnaire score from baseline to the end of study | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Antalya Kepez State Hospital, Antalya, Turkey (Türkiye)